CLINICAL TRIAL: NCT05369819
Title: Effect of Midazolam Premedication on Opioid-induced Mask Ventilation Difficulty During General Anesthesia Induction: A Randomized Clinical Trial
Brief Title: Effect of Midazolam Premedication on Opioid-induced Mask Ventilation Difficulty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karaman Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 08-2021/14
Record Dates: First submitted 2022-04-22; First posted 2022-05-11 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-06

CONDITIONS: Anesthesia Complication
Keywords: premedication; midazolam; opioids; remifentanil; Anesthesia, General
MeSH Terms: interventions — Midazolam; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patients will be unaware of the group assignments and monitored in the reception area by a blinded anesthesiologist who will be in charge of the intervention and the evaluation of anxiety and sedation levels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group M (Experimental): Patients of the Group M will be treated with midazolam premedication.
  Interventions: Drug: Midazolam
- Group S (Placebo Comparator): Group S patients are treated with 3 cc normal saline.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Midazolam — . Patients of the midazolam group will be treated with midazolam premedication (3 cc mixture of 0.035 mg/kg midazolam and normal saline; maximum midazolam dose, 3 mg) intravenously a waiting area 3 minutes before transportation to an operating room
  Other Names: Group M
  Arms: Group M
Drug: Saline — Control group patients are treated with 3 cc normal saline in a waiting area 3 minutes before transportation to an operating room
  Other Names: Group S
  Arms: Group S

SUMMARY:
Mask ventilation has great importance during anesthesia induction because it is the only way to oxygenate patients who have lost consciousness and spontaneous breathing. Opioid-derived drugs used in anesthesia induction may cause difficulty in mask ventilation due to their chest wall rigidity and respiratory depressant effects. Adequate muscle relaxation and depth of anesthesia may assist with mask ventilation. It is known that premedication reduces anxiety and has a relaxing effect on airway muscles. Midazolam is frequently used in premedication because it has a rapid onset of action and does not cause hemodynamic changes. In addition, midazolam may relax the airway by acting directly on the airway smooth muscle and thus facilitate mask ventilation during anesthesia induction. In this study, the investigators will evaluate the effect of midazolam premedication on the mask ventilation after induction with remifentanil.

DETAILED DESCRIPTION:
American Society of Anesthesiologists (ASA) class I and II patients who are admitted to undergoing elective surgery under general anesthesia will be enrolled. Patients in midazolam group (Group M) will be treated with midazolam premedication (3 cc mixture of 0.035 mg/kg midazolam and normal saline; maximum midazolam dose, 3 mg) intravenously in a waiting area 3 minutes before transportation to an operating room, while 3 cc normal saline will be administered to control group (Group S) patients. The difficulty of mask ventilation will be evaluated before the injection of neuromuscular blocking during general anesthetic induction. The anxiety and sedation levels of patients will be estimated before the intervention and before anesthetic induction in an operating room. Remifentanil will be used as an opioid in the induction of the patients. In anesthesia induction, propofol 1.5 mg/kg will be given after remifentanil is infused at a dose of 0.30 µg/kg/min for three minutes. Before the patients were given muscle relaxants, the patients were evaluated with the Warter scale

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) class I and II patients
* Patients who are scheduled for any elective surgery under general anesthesia

Exclusion Criteria:

* age <18 or >60 years
* current cervical spine disease or history of cervical spine surgery;
* morbid obesity (body mass index, ≥35 kg/m2);
* sleep apnea;
* craniofacial anomaly;
* allergic reaction to midazolam and remifentanil
* chronic use of opioid, benzodiazepine, antipsychotic medications
* pregnancy
* presence of muscle weakness or dyspnea

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-01-03 (Actual)

PRIMARY OUTCOMES:
Difficulty of mask ventilation (Warters grading scale 0-10) | During surgery at 30 seconds after loss of consciousness
  The difficulty of mask ventilation will be assessed after 30 seconds from propofol induction (loss of consciousness) with Warter's scale.
  The Warters scale assigns points based on escalating levels of intervention necessary to ventilate the lungs such as the use of an airway device, increased inspiratory pressure, and two-person ventilation, which are all intended to overcome upper airway resistance to ventilation. Additionally, the Warters scale accounts for situations in which a poor quality mask seal inhibits mask ventilation. Thus, in the event that the target tidal volume of 5 ml/kg is not achieved, and the provider is unable to generate a peak inspiratory pressure of >30 cmH20, additional points are assigned. The scale is scored between 0-10 and higher scores indicate worse mask application.

SECONDARY OUTCOMES:
Anxiety level; Numerical Rating Scale(NRS) score (0 - 10) | One minute before the intervention in waiting area, and one minute before the anesthetic induction in operating room
  The NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0 to 10 integers) that best reflects the intensity of their anxiety (0= very calm, 10= very anxious).
Sedation level (Modified Observer's assessment of alertness/sedation (MOAA/S) scale) | One minute before the intervention in waiting area, and one minute before the anesthetic induction in operating room
  Before the intervention in the waiting area, and before the anesthetic induction in the operating room sedation levels were evaluated with MOAA/S scale. The Modified Observer's Assessment of Alertness/Sedation (MOAA/S) Scale was developed to measure the level of alertness in subjects who are sedated. The Modified Observer's Assessment of Alertness and Sedation (MOAA/S) scale is frequently used in sedation-related drug and device studies to assess a subject's level of sedation. The MOAA/S ranges from 0 to 5, with a score of 5 defined as awake or minimally sedated, and a score of 0 defined as general anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Rafet Yarımoglu, MD, Principal Investigator — Karaman Training and Research Hospital
Locations (1):
- Karaman Training and Research Hospital, Karaman, Turkey (Türkiye)